CLINICAL TRIAL: NCT00512031
Title: Characterizing the Effects of PAI-1 Modulation on Human Monocyte Function - The Effect of PAI-1 Post-transcriptional Regulation on Human Monocyte Adhesion
Brief Title: Characterizing PAI-1 Modulation on Monocyte Adhesion
Status: Terminated | Type: Observational
Why Stopped: Investigator left institution
Sponsor: Vanderbilt University (Other)
Responsible Party: Mohan Sathyamoorthy, Vanderbilt University
Other Study IDs: 070079
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; metabolic pathways; monocyte adhesion,
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine how altering the expression of a gene known as PAI-1 may affect the adhesive capacity of cells that play a critical role in the developement of human atherosclerosis.

DETAILED DESCRIPTION:
The principal aim of this study is to determine if molecular regulation of the human gene PAI-1 alters the migratory properties of human myeloid and endothelial cells sufficiently enough to regulate entry and exit from the vascular space. Human monocyte become the key cellular orchestrators of human atherosclerotic plaque. We believe that a "loss" of PAI-1 activity may promote a pro-atherogenic effect in human vasculature thereby defining a novel atheroprotective effect for PAI-1 when expressed at normal levels in humans. By using RNA interference to achieve PAI-1 gene, we hope to elucidate the mechanistic basis of how PAI-1 regulation may affect human migration within the vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* No current or past medical problems

Exclusion Criteria:

* Patients taking prescription drugs (hormonal birth control or herbal supplements may be taken)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Sathyamoorthy, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States